CLINICAL TRIAL: NCT03698331
Title: A Phase 4, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Potential for Clinical Dependence and Withdrawal Symptoms Associated With Valbenazine
Brief Title: The Potential for Clinical Dependence and Withdrawal Symptoms Associated With Valbenazine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBI-98854-TD4001
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Tardive Dyskinesia (TD)
MeSH Terms: conditions — Tardive Dyskinesia | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Valbenazine (Experimental): Valbenazine or placebo oral capsules administered once daily for 7 weeks.
  Interventions: Drug: Valbenazine; Drug: Placebo oral capsule
- Placebo (Placebo Comparator): Placebo oral capsules administered once daily for 7 weeks.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Valbenazine — vesicular monoamine transporter 2 (VMAT2) inhibitor
  Other Names: Ingrezza, NBI-98854
  Arms: Valbenazine
Drug: Placebo oral capsule — non-active dosage form

SUMMARY:
This is a Phase 4, randomized, double-blind, placebo-controlled study to evaluate the potential for clinical dependence and withdrawal symptoms associated with valbenazine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of childbearing potential must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment, and follow-up periods of the study.
2. Have one of the following clinical diagnoses for at least 3 months before screening: Schizophrenia, Schizoaffective Disorder, or Mood Disorder
3. Have a clinical diagnosis of neuroleptic-induced TD for at least 3 months before screening.
4. Be on stable doses if using maintenance medication(s) for schizophrenia or schizoaffective disorder, or mood disorder. Subjects with bipolar disorder must be on stable doses of a mood stabilizer.
5. Be in general good health.
6. Have adequate hearing, vision, and language skills to perform the procedures specified in the protocol.

Exclusion Criteria:

1. Have an active, clinically significant unstable medical condition within 1 month before screening.
2. Have a known history of substance (drug) dependence, or substance or alcohol abuse.
3. Have a significant risk of suicidal or violent behavior.
4. Have a known history of neuroleptic malignant syndrome.
5. Have a known history of long QT syndrome or cardiac arrhythmia.
6. Have a cancer diagnosis within 3 years prior to screening (some exceptions allowed).
7. Have ever taken valbenazine (INGREZZA or NBI-98854) or participated in a valbenazine clinical study.
8. Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study.
9. Have a blood loss ≥550 mL or donated blood within 30 days prior to Baseline.
10. Have an allergy, hypersensitivity, or intolerance to VMAT2 inhibitors (eg, tetrabenazine, deutetrabenazine).
11. Are currently pregnant or breastfeeding.
12. Have HIV or hepatitis B.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Chief Medical Officer
Locations (15):
- United States (14):
  - Neurocrine Clinical Site, Anaheim, California
  - Neurocrine Clinical Site, Glendale, California
  - Neurocrine Clinical Site, Norwalk, California
  - Neurocrine Clinical Site, Oceanside, California
  - Neurocrine Clinical Site, San Bernardino, California
  - Neurocrine Clinical Site, Hialeah, Florida
  - Neurocrine Clinical Site, Honolulu, Hawaii
  - Neurocrine Clinical Site, Fort Wayne, Indiana
  - Neurocrine Clinical Site, Ann Arbor, Michigan
  - Neurocrine Clinical Site, Beechwood, Ohio
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, Scranton, Pennsylvania
  - Neurocrine Clinical Site, DeSoto, Texas
  - Neurocrine Clinical Site, Irving, Texas
- Neurocrine Clinical Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Valbenazine/Placebo: Valbenazine administered once daily for 4 weeks, followed by placebo administered once daily for 3 weeks.
- Placebo/Placebo: Placebo administered once daily for 7 weeks.
Period: Overall Study
Arm/Group | Valbenazine/Placebo | Placebo/Placebo
Started | 44 | 45
Entered Withdrawal Period | 42 | 39
Completed | 40 | 39
Not Completed | 4 | 6
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Non-compliance with study drug | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valbenazine/Placebo | Placebo/Placebo | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (7.5) | 53.6 (9.5) | 54.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 25 | 27 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 17 | 36
  Not Hispanic or Latino | 25 | 28 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 19 | 32
  White | 30 | 25 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants With Withdrawal-Emergent Adverse Events
Description: A withdrawal-emergent adverse event is an adverse event that begins during the Withdrawal Period.
Time Frame: 3 weeks
Population: Dependence and Withdrawal Analysis Set, which includes all participants who were randomized, took at least one dose of study drug, and entered the Withdrawal Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Valbenazine/Placebo | Placebo/Placebo
Number analyzed (Participants) | 42 | 39
Participants | 9 | 13

2. Secondary Outcome: Participants Who Experience Worsening of Symptoms as Measured by the Physician Withdrawal Checklist-20 (PWC-20)
Description: The PWC-20 is a validated 20-item physician-rated survey that assesses the severity of potential symptoms of withdrawal. Items are rated on a scale from 0 to 3, with total scores ranging from 0 to 60. Worsening of symptoms is defined by 5 new symptoms of moderate or severe degree or a worsening of symptoms by 2 points on the PWC-20 scale during Weeks 5 to 7 compared with Week 4. Note: a 2-point worsening from 0 (none) at Week 4 to 2 (moderate) post-Week 4 is counted as a worsening of symptoms.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Valbenazine/Placebo | Placebo/Placebo
Number analyzed (Participants) | 42 | 39
Participants | 9 | 3

3. Secondary Outcome: Absolute Worst Total Score as Measured by the Physician Withdrawal Checklist-20 (PWC-20)
Description: The PWC-20 is a validated 20-item physician-rated survey that assesses the severity of potential symptoms of withdrawal. Items are rated on a scale from 0 to 3, with total scores ranging from 0 to 60. Larger values indicate more severe symptoms. Rickels et al (J Clin Psychopharmacol 2008) cites PWC-20 mean scores associated with withdrawal in the range of 15 to 24.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valbenazine/Placebo | Placebo/Placebo
Number analyzed (Participants) | 42 | 39
score on a scale
  Mean absolute score at baseline | 4.6 (5.0) | 3.9 (4.5)
  Mean absolute score at withdrawal baseline | 3.8 (3.7) | 3.1 (3.8)
  Mean absolute worst total score | 5.6 (5.3) | 3.3 (2.6)

4. Secondary Outcome: Severity of Withdrawal Symptoms as Measured by the Change From Withdrawal Baseline (Week 4) to Week 7 in the Modified Cocaine Selective Severity Assessment (mCSSA)
Description: The mCSSA is an 18-item survey based on symptoms commonly associated with early cocaine abstinence, including depression, fatigue, anhedonia, anxiety, irritability, sleep disturbance, and inability to concentrate. Items are rated on scales of 0 to 7 or 0 to 8, with separate scale descriptions for each item. Larger values indicate more severe symptoms. The scale has been modified to be specific to study drug (valbenazine or placebo) instead of cocaine.
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valbenazine/Placebo | Placebo/Placebo
Number analyzed (Participants) | 42 | 39
score on a scale | 1.9 (4.1) | 0.5 (3.2)

5. Secondary Outcome: Overall Improvement From Baseline of TD Symptoms as Measured by the Clinical Global Impression-Tardive Dyskinesia-Improvement (CGI-TD-I) Score
Description: The CGI-TD-I scale is a 7-point scale (range; 1=very much improved to 7=very much worse) used to assess overall improvement in TD symptoms since the initiation of study drug dosing.
Time Frame: Baseline, Week 4, Week 7
Population: Efficacy analysis set was defined as all participants who were randomized to a treatment group, took at least one dose of study drug, and had a CGI-TD-I assessment at Week 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valbenazine/Placebo | Placebo/Placebo
Number analyzed (Participants) | 41 | 40
score on a scale
  End of Week 4 | 3.2 (0.8) | 3.4 (0.7)
  End of Week 7: number analyzed (Participants) | 40 | 39
  End of Week 7 | 3.0 (0.7) | 3.0 (0.8)

6. Secondary Outcome: Change in Severity of TD Symptoms as Measured by Change From Baseline in the Clinical Global Impression-Tardive Dyskinesia-Severity (CGI-TD-S) Scale
Description: The CGI-TD-S scale is a 7-point scale (range; 1=normal, not at all ill to 7=among the most extremely ill patient) used to assess the overall global severity of TD.
Time Frame: Baseline, Week 4, Week 7
Population: Efficacy analysis set was defined as all participants who were randomized to a treatment group, took at least one dose of study drug, and had a CGI-TD-S assessment at Week 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valbenazine/Placebo | Placebo/Placebo
Number analyzed (Participants) | 41 | 40
score on a scale
  End of Week 4 | -0.3 (0.7) | -0.2 (0.6)
  End of Week 5: number analyzed (Participants) | 40 | 38
  End of Week 5 | -0.3 (0.6) | -0.3 (0.6)
  End of Week 6: number analyzed (Participants) | 40 | 39
  End of Week 6 | -0.4 (0.5) | -0.5 (0.6)
  End of Week 7: number analyzed (Participants) | 40 | 39
  End of Week 7 | -0.4 (0.5) | -0.5 (0.6)

ADVERSE EVENTS:
Time Frame: Up to 7 weeks
Arm/Group | Valbenazine/Placebo | Placebo/Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/44 | 1/45
Other Adverse Events (participants affected / at risk) | 12/44 | 19/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine/Placebo (N=44) | Placebo/Placebo (N=45)
Schizoaffective disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine/Placebo (N=44) | Placebo/Placebo (N=45)
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 5
Somnolence (Nervous system disorders) | 2 | 1
Dry eye (Eye disorders) | 2 | 1
Fatigue (General disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 4
Anxiety (Psychiatric disorders) | 1 | 2
Hypertension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT03698331/SAP_000.pdf
  • Study Protocol (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT03698331/Prot_001.pdf